CLINICAL TRIAL: NCT00449956
Title: Multicenter, Double-Blind, Active Comparator-controlled Study to Evaluate the Safety and Efficacy of MK0507A in Patients With Glaucoma and Ocular Hypertension Who Are Inadequately Controlled on Beta-Blockers
Brief Title: MK0507A Clinical Study in Patients With Glaucoma and Ocular Hypertension (0507A-149)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0507A-149; MK0507A-149; 2007_011
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Results first posted 2009-05-29 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): combination of dorzolamide hydrochloride and timolol maleate
  Interventions: Drug: dorzolamide hydrochloride (+) timolol maleate
- 2 (Active Comparator): Concomitant use of dorzolamide hydrochloride and timolol maleate
  Interventions: Drug: Comparator: timolol maleate; Drug: Comparator: dorzolamide hydrochloride
- 3 (Active Comparator): timolol maleate
  Interventions: Drug: Comparator: timolol maleate

INTERVENTIONS:
Drug: dorzolamide hydrochloride (+) timolol maleate — Dorzolamide hydrochloride 1% + timolol 0.5%, 8-week
  Arms: 1
Drug: Comparator: timolol maleate — timolol maleate 0.5%, 8-week
  Arms: 2; 3
Drug: Comparator: dorzolamide hydrochloride — dorzolamide hydrochloride 1%, 8-week
  Arms: 2

SUMMARY:
The clinical study compares safety and efficacy of MK0507A (dorzolamide 1.0% / timolol 0.5%) with 1) timolol 0.5% and with 2) concomitant therapy with dorzolamide 1.0% / timolol 0.5% in patients with glaucoma and ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma and ocular hypertension

Exclusion Criteria:

* History of ocular surgery within 3 months
* Administration contradiction to timolol and dorzolamide

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2007-03-12 (Actual); Primary Completion 2008-02-16 (Actual); Study Completion 2008-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kitazawa Y, Araie M; Research Group on MK-0507A. [Double-masked, phase III comparative study of the combination ophthalmic solution of the 1% dorzolamide hydrochloride/0.5% timolol maleate (MK-0507A) in patients with glaucoma and ocular hypertension]. Nippon Ganka Gakkai Zasshi. 2011 Jun;115(6):495-507. Japanese. PMID 21735753

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III.
  Studied period: April 9, 2007 (date study therapy started for the first subject) to February 16, 2008 (the last subject's last visit stipulated in study protocol). Study was conducted at 67 clinical sites.
Pre-assignment Details: Outpatients with primary open angle glaucoma (broad definition) and/or ocular hypertension received 4-week timolol 0.5% monotherapy in the wash-out period before the study randomization.
Groups:
- MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination): MK0507A (Dorzolamide 1.0% / Timolol 0.5% combination), one drop per dose twice daily to the study eye.
- Timolol 0.5%: Timolol 0.5%, one drop per dose twice daily to the study eye.
- Concomitant (Dorzolamide 1.0% / Timolol 0.5%): Concomitant (Dorzolamide 1.0%, one drop per dose three times daily to the study eye / Timolol 0.5%, one drop per dose twice daily to the study eye).
Period: Overall Study
Arm/Group | MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) | Timolol 0.5% | Concomitant (Dorzolamide 1.0% / Timolol 0.5%)
Started | 189 | 92 | 193
Completed | 179 | 88 | 184
Not Completed | 10 | 4 | 9
Not completed — Adverse Event | 7 | 1 | 6
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) | Timolol 0.5% | Concomitant (Dorzolamide 1.0% / Timolol 0.5%) | Total
Number analyzed (Participants) | 189 | 92 | 193 | 474
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (10.8) | 61.3 (11.6) | 62.3 (12.7) | 62.4 (11.7)
Age, Customized [Number; unit: participants]
  <65 years | 92 | 50 | 102 | 244
  >=65 years | 97 | 42 | 91 | 230
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 43 | 98 | 245
  Male | 85 | 49 | 95 | 229
Diagnosis [Number; unit: participants]
  Open-angle glaucoma | 107 | 51 | 90 | 248
  Normal-tension glaucoma | 8 | 6 | 4 | 18
  Ocular hypertension | 74 | 35 | 99 | 208
Intraocular pressure (IOP) at Hour 2 [Mean (Standard Deviation); unit: mmHg] | 20.54 (2.07) | 20.23 (1.85) | 20.38 (2.31) | 20.42 (2.13)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) From Baseline at 8 Weeks
Description: Change from baseline to 8 weeks in Intraocular Pressure (IOP) assessed 2 hours after ocular instillation (at Hour 2)
Time Frame: 8 weeks
Population: Last observed value during the 8-week treatment period was used in the Full Analysis Set (FAS).
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) | Timolol 0.5% | Concomitant (Dorzolamide 1.0% / Timolol 0.5%)
Number analyzed (Participants) | 185 | 90 | 188
mmHg | -2.50 [-2.86 to -2.15] | -1.82 [-2.33 to -1.31] | -2.78 [-3.13 to -2.43]
Statistical Analysis 1: Comparison: MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) vs Timolol 0.5%; Test type: Superiority or Other; Mean Difference (Final Values) = -0.68, 95% CI [-1.30 to -0.06] — An analysis of covariance model with a factor for treatment and time-matched baseline as a covariate was used to compute 95% confidence intervals
Statistical Analysis 2: Comparison: MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) vs Concomitant (Dorzolamide 1.0% / Timolol 0.5%); Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 1.2 mmHg; Mean Difference (Final Values) = 0.28, 95% CI [-0.22 to 0.78] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percent Change From Baseline in Intraocular Pressure (IOP) at 8 Weeks
Description: Percent Change from baseline to 8 weeks in Intraocular Pressure (IOP) assessed 2 hours after ocular instillation (at Hour 2)
Time Frame: 8 Weeks
Population: Last observed value during the 8-week treatment period was used in the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) | Timolol 0.5% | Concomitant (Dorzolamide 1.0% / Timolol 0.5%)
Number analyzed (Participants) | 185 | 90 | 188
Percent Change | -11.99 [-13.69 to -10.28] | -8.74 [-11.18 to -6.30] | -13.46 [-15.15 to -11.77]

3. Secondary Outcome: Percent Change From Baseline in Outflow Pressure Reduction Rate at 8 Weeks
Description: Percent Change from baseline to 8 weeks in Outflow Pressure Reduction Rate assessed 2 hours after ocular instillation (at Hour 2)
Time Frame: 8 weeks
Population: Last observed value during the 8-week treatment period was used in the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) | Timolol 0.5% | Concomitant (Dorzolamide 1.0% / Timolol 0.5%)
Number analyzed (Participants) | 185 | 90 | 188
Percent Change | 23.47 [20.07 to 26.88] | 17.17 [12.29 to 22.05] | 26.75 [23.37 to 30.12]

ADVERSE EVENTS:
Arm/Group | MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) | Timolol 0.5% | Concomitant (Dorzolamide 1.0% / Timolol 0.5%)
Serious Adverse Events (participants affected / at risk) | 2 | 1 | 0
Other Adverse Events (participants affected / at risk) | 36 | 12 | 40
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) | Timolol 0.5% | Concomitant (Dorzolamide 1.0% / Timolol 0.5%)
Arteriosclerosis obliterans (Vascular disorders) | 1/189 | 0/92 | 0/193
Forearm fracture (Injury, poisoning and procedural complications) | 0/189 | 1/92 | 0/193
Cerebral infarction (Nervous system disorders) | 1/189 | 0/92 | 0/193
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | MK0507A (Dorzolamide 1.0% / Timolol 0.5% Combination) | Timolol 0.5% | Concomitant (Dorzolamide 1.0% / Timolol 0.5%)
Conjunctival hyperaemia (Eye disorders) | 3/189 | 1/92 | 4/193
Corneal epithelium defect (Eye disorders) | 2/189 | 2/92 | 5/193
Punctate keratitis (Eye disorders) | 3/189 | 0/92 | 6/193
Instillation site irritation (General disorders) | 13/189 | 0/92 | 7/193
Nasopharyngitis (Infections and infestations) | 5/189 | 3/92 | 8/193
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/189 | 1/92 | 4/193
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0/189 | 2/92 | 0/193
Headache (Nervous system disorders) | 4/189 | 0/92 | 0/193
Alanine aminotransferase increased (Investigations) | 4/189 | 2/91 | 5/193
Glucose urine present (Investigations) | 5/189 | 1/91 | 9/193
Blood urine present (Investigations) | 3/198 | 3/91 | 0/193

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.